CLINICAL TRIAL: NCT00729027
Title: A Multicenter, Double-blind, Randomized, 12-month, Placebo-controlled Study to Evaluate the Lipid-lowering Effect, Safety and Tolerability of AVE5530 25 mg/Day and 50mg/Day When Added to Ongoing Stable Statin Therapy (HMG-CoA Reductase Inhibitors) in Patients With Primary Hypercholesterolemia
Brief Title: Evaluation of Safety and Efficacy of AVE5530 as add-on to Ongoing Statins in Patients With Primary Hypercholesterolemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: AVE5530 in hypercholesterolemia was stopped due to insufficient efficacy
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC6910; EudraCT: 2008-001550
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 25 mg/day AVE5530 (Experimental)
  Interventions: Drug: 25 mg/day AVE5530
- 50 mg/day AVE5530 (Experimental)
  Interventions: Drug: 50 mg/day AVE5530
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 25 mg/day AVE5530 — * one tablet in the evening with dinner
  * in addition to statin treatment (HMG-CoA Reductase Inhibitors)
  Arms: 25 mg/day AVE5530
Drug: 50 mg/day AVE5530 — * one tablet in the evening with dinner
  * in addition to statin treatment (HMG-CoA Reductase Inhibitors)
  Arms: 50 mg/day AVE5530
Drug: placebo — * one tablet in the evening with dinner
  * in addition to statin treatment (HMG-CoA Reductase Inhibitors)
  Arms: Placebo

SUMMARY:
The present study is assessing the efficacy and safety of AVE5530 (25 mg and 50 mg) in add-on to ongoing statin treatment in a double-blind manner in comparison with placebo, in the management of patients with primary hypercholesterolemia considered as inadequately controlled despite their ongoing statin treatment.

The main objective is to evaluate the effects of the association AVE5530+statin on LDL-C level reduction after 12 weeks of treatment. The effects of AVE5530 on other lipid parameters will be assessed as secondary objectives.

DETAILED DESCRIPTION:
The two doses of AVE5530 tested in this study are 25 mg and 50 mg taken in the evening, with dinner dosing. The study will include a screening phase up to 2 weeks, a double-blind treatment period of at least 12 months and can be variably extended up to approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults with cholesterol levels not controlled on ongoing stable statin treatment

Exclusion Criteria:

* LDL-C levels > 250 mg/dL (6.48 mmol/L)
* Triglycerides >350 mg/dL (3.95 mmol/L)
* Conditions / situations such as:

  * presence of any clinically significant uncontrolled endocrine disease known to influence lipids levels
  * Active liver disease
  * Recent history of congestive heart failure , of unstable angina pectoris, myocardial infarction, coronary bypass surgery or angioplasty, or Unstable or severe peripheral artery disease
  * Positive test for Hepatitis B surface antigen and/or Hepatitis C antibody or Known to be Human Immunodeficient Virus (HIV) positive
* Pregnant or breast-feeding women,
* Women of childbearing potential not protected by effective contraceptive method of birth control (including oral contraceptives) and/or who are unwilling or unable to be tested for pregnancy prior to exposure to the Investigational Product

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in calculated LDL-C | At week 12

SECONDARY OUTCOMES:
Percent change from baseline in calculated LDL-C | At 6 months and 12 months
Percent change from baseline in Total-Cholesterol and Apo-B | At 12 weeks, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mats ERICKSSON, MD, Principal Investigator — Department of Endocrinology, Metabolism and Diabetes, Karolinska University Hospital, Huddinge, Sweden
Locations (16):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden